#### RESEARCH PROTOCOL

| Date | 5-15-19 |
|---|---|
| Title | Female Patient Preferences regarding Physician Gender; is there a |
| | difference? A National Survey |
| Principal Investigator | Rachel Pauls, MD |
| Sub-Investigators | Tiffanie Tam, MD; Austin Hill, MD |
| Research Specialist | Eunsun Yook, MS |
| Department | Female Pelvic Medicine and Reproductive Surgery |
| Hatton # | 18-113 |

| IRB Review Type: | Exempt | Expedited | Full Board |
|------------------|--------|-----------|------------|
|------------------|--------|-----------|------------|

# **Purpose of Study**

- Primary Aim: To describe female patient preferences when choosing their OB/GYN and other providers.
- Secondary Aim:
- To assess these preferences based on patient demographic factors as well as physician specialty.
- To assess qualities which are most important to female patients when choosing a physician.

### **Hypothesis or Research Question**

 We hypothesize that females are not more likely to choose a female physician, in particular for their OB/GYN care

#### **Background**

In 2017, the AAMC published that the number of women accepted into US medical schools increased by 3.2% and the female students represented 50.7% of the new enrollees [1]. This represents a dramatic increase in female trainees over the past decade. Furthermore, the American College of Obstetricians and Gynecologists (ACOG) published that as of 2009, 79.7% of the Obstetrics and Gynecology residents were female [2]. This gender disparity could be related to perceived limitations in practice, leading to fewer males selecting this specialty.

Nevertheless, it is not clear that females have strong preferences regarding gender. One study revealed that 34% of women preferred females because they were "more comfortable" and "easier to talk to", 58% had no preference and only 7% preferred male providers because they were "more gentle" and "more compassionate" [3, 4]. Another study reported that of the qualities when choosing an OB/GYN, it was experience, knowledge and ability that were what patients looked for over 15.7% reporting gender was a role in choice of physician [3].

The overall conclusion drawn from these studies was that female physician choice is less based on gender preference and more on characteristic qualities [2-5]. However, women aged ≤25

preferred a female physician versus women 42.4 years and older [3, 7]. This data collected was published more than 10 years ago. Given the striking decline in male providers selecting OB/GYN in more recent years, it is critical to characterize patient preferences in the current environment. We hope to better understand the influence of bias on physician gender in present day.

#### **Research Plan**

## Study Design

This will be a cross sectional survey conducted via an online server

## **Setting for the study**

The study will be conducted on an online platform distributed across the United States by the aid of Survey Monkey

### Participants

- Study population: All women between 18 and 80 years of age residing in the USA
- o Inclusion/Exclusion criteria:
  - Inclusion
    - Females between 18 and 80 years of age (this will be selected) during the target population inquiry within the survey limits)
  - **Exclusion** 
    - Unwillingness to participate in the study
    - Lack of access to the internet
    - Non-English speaking
  - Sample size
    - We hope to gather 1000 responses from females across the U.S.
    - SurveyMonkey® will use their databank to recruit enough panelists for obtaining 1000 responses.

#### **Data Collection**

- Primary Outcome:
  - Describe female population preferences based on physician gender
- **Secondary Outcomes:** 
  - Describe qualities that female patients use to choose physicians
  - Describe if physician specialty plays a role in choice
  - Describe demographic factors that may predict patient preferences, such as age, race, socioeconomic factors
- General demographic data:
  - Age, ethnicity, religion, parity, income level, education level, marital status, medical insurance status, number of regularly seen providers
- Intervention or experimental aspect of the study
  - Procedure

 Study group will be surveyed online using Survey Monkey using the Physician Preference Survey designed by the investigators.

#### **Statistical Analysis**

• Demographic data will be described using frequency (percentage). The association between the preference on physician gender and demographic factors will be assessed by Pearson's chi-square test. Logistic regression will be used to investigate whether the preference on physician gender can be predicted based on a demographic factor(s).

#### **Ethical Considerations**

#### • Informed consent

 By completing the survey patients will consent to participating in the study. A waiver of documentation of informed consent will be requested.

### **Privacy information**

- Because this is an online anonymous conducted survey, there will be no available identifying information.
- Participants however, will be logged in the Excel spreadsheet and assigned a Subject ID number. Each participant will be assigned the next available Subject ID number. Once each Subject ID number has been assigned, it will not be reassigned. The Excel spreadsheet will be stored on a password protected, encrypted TriHealth computer for ten years following study closure, and then purged.

# Cost/Budget

| cost baubet | | | |
|---|---|---|---|
| Item | Qty | Cost per Item | Total |
| Survey Monkey Responses needed | 1000 | \$2.50 | \$2500.00 |
| Unlimited questions with Advantage plan | 20 | 0 | 0 |
| Survey Monkey Advantage Plan | 1 | Paid by Hatton<br>Account | 0 |
| Total | | | \$2500.00 |

| Estimated Period of Time to Complete Study | |
|---|---|
| When will study begin? | January 15 <sup>th</sup> , 2019 |
| Protocol Development<br>Completed | November 30 <sup>rd</sup> , 2018 |

| Admin Review Time | 2 weeks |
|---|---|
| IRB Approval | December 18, 2018 |
| Data collection | Subjects to be enrolled starting January 15 <sup>th</sup> , 2019 |
| Data analysis | February 2019 |

#### When and how will results be disseminated?

Submit for abstract presentation at national/international meeting and publication

#### References

- [1] "More Women Than Men Enrolled in U.S. Medical Schools in 2017." AAMCNews, 18 Dec. 2017, news.aamc.org/press-releases/article/applicant-enrollment-2017/
- [2] Rayburn, William F. "Women's Health Care Physicians." The Obstetrician- Gynecologist Workforce in the United States: Facts, Figures, and Implications 2017. ACOG, www.acog.org/Clinical-Guidance-and-Publications/The-Ob-Gyn-Workforce/The-Obstetrician-Gynecologist-Workforce-in-the-United-States.
- [3] Johnson, Amy M., et al. "Do Women Prefer Care From Female or Male Obstetrician-Gynecologists? A Study of Patient Gender Preference." The Journal of the American Osteopathic Association, American Osteopathic Association, 1 Aug. 2005, jaoa.org/article.aspx?articleid=2093065
- [4] Howell, Elizabeth, and John Concato. "Do Women Prefer Female Obstetricians?" Obstetrics & Gynecology, vol. 100, no. 4, 2002, p. 828., doi:10.1097/00006250-200210000-00035.
- [5] Haar E, Halitsky V, Stricker G. Factors related to the preference for a female gynecologist. *Med Care.* 1975;13:782-790.
- [6] Fisher WA, Bryan A, Dervaitis KL, Silcox J, Kohn H. It aint' necessarily so: most women do no strongly prefer female obstetrician-gynaecologists. J obstet Gynaecol Can. 2002;24:885-888.
- [7] Yanikkerem, Emre, et al. "Women's Attitudes and Expectations Regarding Gynaecological Examination." Current Neurology and Neuroscience Reports., U.S. National Library of Medicine, Oct. 2009, www.ncbi.nlm.nih.gov/pmc/articles/PMC2801597/.